CLINICAL TRIAL: NCT00872794
Title: Prospective Single-centre, Uncontrolled, Post Marketing Surveillance Study to Monitor the Long-term Performance of the DePuy ASR™ Hip in Subjects With Suitable Indications for a Primary Resurfacing Hip Arthroplasty
Brief Title: A Single Centre Study to Assess the Long-term Performance of the DePuy ASR™ System in Primary Hip Resurfacing Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: DePuy discontinued this product in 4Q 2009.At the time of this decision DePuy reviewed all clinical studies for this product and decided to close this Study.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT03/29
Record Dates: First submitted 2009-03-19; First posted 2009-03-31 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Conservative; Metal on Metal; Resurfacing
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DePuy ASR Hip System (Other): A metal-on-metal bearing surface replacement system for use in resurfacing hip arthroplasty.
  Interventions: Device: DePuy ASR™ Hip System

INTERVENTIONS:
Device: DePuy ASR™ Hip System — A metal-on-metal bearing surface replacement system for use in resurfacing hip arthroplasty.

SUMMARY:
The purpose of this study is to monitor the performance and determine the metal ion release of the DePuy ASR™ System in the treatment of patients with hip joint disease requiring hip resurfacing surgery. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments. A subset of patients will also have blood samples taken at regular intervals to allow the metal ion levels to be determined and undergo scans to allow the bone mineral density of the bone surrounding the implant to be monitored.

DePuy decided to close this Study in 4Q 2009. The Study was terminated with effect from November 2010 to allow for the completion of the 5 year follow up assessments.

Please note that subsequent to this decision DePuy voluntarily recalled the ASR products on 24 August 2010. Additional information regarding this voluntary recall and the follow-up of patients affected by the recall can be found at the following links http://www.mhra.gov.uk/Publications/Safetywarnings/MedicalDeviceAlerts/CON079157 and http://www.depuy.com/countries_list.

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects, aged between 18 and 65 years inclusive.

ii) Subjects with current indications for standard MoM hip resurfacing arthroplasty suitable for cementless fixation in the acetabulum. These include pain, deformity, and loss of function, which are not responsive to medical treatment.

iii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iv) Subjects, who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.

ii) Subjects with proven significant osteoporosis and poor bone quality.

iii) Subjects with compromised renal function.

iv) Subjects with proven metal sensitivity.

v) Subjects with infectious, highly communicable diseases, which may limit follow-up i.e. Active tuberculosis, hepatitis, immuno-compromised conditions, etc.

vi) Women who are pregnant.

vii) Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.

viii) Subjects who have participated in a clinical study with an investigational product in the last 6 month(s).

ix) Subjects who are currently, or have been in the last 12 months, participating in a clinical study which involves exposure to ionising radiation.

x) Subjects who are currently involved in any injury litigation claims.

Additional Exclusion Criteria for Subjects Undergoing Blood Analysis

1. Subjects who currently have other metallic foreign bodies including trauma products and joint arthroplasties unless known to be pure titanium, titanium alloy.
2. Subjects who, in the opinion of the investigator, will possibly require a separate joint replacement operation within the next two years, including revision operations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship at two years | 2 years

SECONDARY OUTCOMES:
UCLA Activity Score | Annually
WOMAC Score | Annually
Activity Assessment. | Annually
Kaplan-Meier survivorship calculation | Annually
Harris Hip Score | pre-discharge, 3mths, 1yr, 2yrs, 5yrs,10yrs and 15yrs post-surgery
Radiographic analysis | pre-discharge, 3mths, 1yr, 2yrs, 5yrs,10yrs and 15yrs post-surgery
Metal ion analysis in whole blood | 3mths, 6mths, 1yr, 2yrs and 5 yrs post-surgery
Bone mineral density (DEXA) | 3mths, 1yr, 2yrs and 5 yrs post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- St Augustine's Hospital, Durban, South Africa